CLINICAL TRIAL: NCT03964545
Title: Proof-of-concept and Validity of Amygdala-neurofeedback in Adolescent Patients With Emotion Dysregulation
Brief Title: Neurofeedback in Adolescents With Emotion Dysregulation
Acronym: EFPTest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Christian Paret, Principal Investigator, Central Institute of Mental Health, Mannheim
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-519N-MA
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Emotional Disturbances
Keywords: Borderline; Post-traumatic stress; Neurofeedback; Amygdala; Emotion regulation
MeSH Terms: conditions — Affective Symptoms; Emotional Regulation | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFP neurofeedback (Experimental): Ten sessions of EFP neurofeedback training. EEG is picked up with scalp electrodes, processed in real-time and returned to patients. One session lasts 30 min.
  Interventions: Behavioral: neurofeedback
- Treatment as usual (No Intervention): Like patients from the treatment arm, these patients are on current residential treatment.

INTERVENTIONS:
Behavioral: neurofeedback — Patients are instructed to reduce amygdala activation by means of down-regulating the EFP. An auditory feedback interface is used with the instruction to down-regulate volume of a jingle, reflecting intensity of EFP.
  Arms: EFP neurofeedback

SUMMARY:
A treatment to improve emotion regulation is tested in young patients with trauma-related mental disorder. The Electrical FingerPrint (EFP) from the amygdala is used for presenting patients with feedback (i.e. neurofeedback) from the amygdala, a brain region which plays a critical role in emotion and mental disorder. Via feedback, patients learn to self-regulate the neural circuit of emotion.

DETAILED DESCRIPTION:
The study tests a neurofeedback treatment for emotion regulation training in adolescent patients suffering from emotional disturbances, indicated by diagnosis with borderline personality disorder (BPD) and/or post-traumatic stress disorder (PTSD), using innovative Electric Finger-Print (EFP) technology. With neurofeedback, patients can learn to regulate brain activation from emotion brain circuit. The technique allows neurofeedback training of sub-cortical brain activation outside the brain scanner, using an electroencephalography (EEG) surrogate of amygdala activation. The novel approach combines the advantages of functional magnetic resonance imaging (fMRI, i.e. high spatial resolution) and EEG (high scalability). EFP allows the probing of deep brain signals with scalp-electrodes, thus bridging a technological gap in neurofeedback training. The developers used EEG feature extraction and machine learning to receive model coefficients (i.e. the EFP) predicting amygdala BOLD activation based on EEG-channel activity (see Citations in this registration).

Participation in this trial is offered to patients who receive residential treatment at the adolescence center of the Central Institute of Mental Health (Mannheim, Germany) to obtain proof-of-concept in this special population, and to show potential value of adjuvant neurofeedback treatment. Patients in the treatment group receive 10 neurofeedback sessions within 5 weeks. Transfer is assessed with neural and questionnaire measures afterwards. A treatment-as-usual (TAU) control group does not receive the neurofeedback. We expect to replicate correlation of EFP with the blood oxygenation level dependent (BOLD) signal from the amygdala, which is tested via simultaneous fMRI-EEG data acquisition post-treatment. Additionally, we assume improved amygdala-BOLD regulation in an fMRI neurofeedback test.

This study aims to extend proof-of-concept of EFP neurofeedback to an adolescent population suffering from severe emotional disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Female patients will be included with four or more BPD and/or PTSD criteria (DSM-5)
* Willingness to participate in the study
* On residential treatment at adolescence center (Central Institute of Mental Health) throughout the study, including assessment of transfer.

Exclusion Criteria:

* General Pharmacological therapy with benzodiazepines
* Substance use
* Pregnancy
* Eplilepsy, traumatic brain injury, brain tumor or otherwise severe neurological or medical history
* BMI > 16.5
* Non-removable electrical implants
* Non-removable ferrous metal implants Permanent make-up and tattoos
* Claustrophobia

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Amygdala self-regulation | Change from baseline to 5 weeks
  Amygdala BOLD regulation is assessed in a transfer task. Transfer task: Two 60s-blocks of BOLD fMRI neurofeedback (visual thermometer) with instruction to down-regulate.

SECONDARY OUTCOMES:
Alexithymia | Change from baseline to 5 weeks
  Impaired cognitive processing of emotion, assessed via questionnaire TAS-26, score range: 0-130 (higher score indicates higher alexithymia)

CONTACTS AND LOCATIONS:
Overall Officials: Paret, Principal Investigator — Central Institute of Mental Health
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keynan JN, Cohen A, Jackont G, Green N, Goldway N, Davidov A, Meir-Hasson Y, Raz G, Intrator N, Fruchter E, Ginat K, Laska E, Cavazza M, Hendler T. Electrical fingerprint of the amygdala guides neurofeedback training for stress resilience. Nat Hum Behav. 2019 Jan;3(1):63-73. doi: 10.1038/s41562-018-0484-3. Epub 2018 Dec 10. PMID 30932053
- [Background] Keynan JN, Meir-Hasson Y, Gilam G, Cohen A, Jackont G, Kinreich S, Ikar L, Or-Borichev A, Etkin A, Gyurak A, Klovatch I, Intrator N, Hendler T. Limbic Activity Modulation Guided by Functional Magnetic Resonance Imaging-Inspired Electroencephalography Improves Implicit Emotion Regulation. Biol Psychiatry. 2016 Sep 15;80(6):490-496. doi: 10.1016/j.biopsych.2015.12.024. Epub 2016 Jan 6. PMID 26996601
- [Background] Meir-Hasson Y, Keynan JN, Kinreich S, Jackont G, Cohen A, Podlipsky-Klovatch I, Hendler T, Intrator N. One-Class FMRI-Inspired EEG Model for Self-Regulation Training. PLoS One. 2016 May 10;11(5):e0154968. doi: 10.1371/journal.pone.0154968. eCollection 2016. PMID 27163677
- [Background] Paret C, Kluetsch R, Zaehringer J, Ruf M, Demirakca T, Bohus M, Ende G, Schmahl C. Alterations of amygdala-prefrontal connectivity with real-time fMRI neurofeedback in BPD patients. Soc Cogn Affect Neurosci. 2016 Jun;11(6):952-60. doi: 10.1093/scan/nsw016. Epub 2016 Feb 1. PMID 26833918
- [Background] Nicholson AA, Rabellino D, Densmore M, Frewen PA, Paret C, Kluetsch R, Schmahl C, Theberge J, Neufeld RW, McKinnon MC, Reiss J, Jetly R, Lanius RA. The neurobiology of emotion regulation in posttraumatic stress disorder: Amygdala downregulation via real-time fMRI neurofeedback. Hum Brain Mapp. 2017 Jan;38(1):541-560. doi: 10.1002/hbm.23402. Epub 2016 Sep 20. PMID 27647695
- [Background] Lubianiker N, Goldway N, Fruchtman-Steinbok T, Paret C, Keynan JN, Singer N, Cohen A, Kadosh KC, Linden DEJ, Hendler T. Process-based framework for precise neuromodulation. Nat Hum Behav. 2019 May;3(5):436-445. doi: 10.1038/s41562-019-0573-y. Epub 2019 Apr 15. PMID 30988481
- See also: Parallel OSF registration — https://osf.io/6zds5